CLINICAL TRIAL: NCT00292331
Title: A Randomized Trial of Endoscopic Treatment of Acute Gastric Variceal Hemorrhage: N-Butyl-2-Cyanoacrylate Injection Versus Band Ligation
Brief Title: N-Butyl-2-Cyanoacrylate Injection Versus Band Ligation for Gastric Variceal Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGH-88-B251
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2006-02-15 (Estimated); Status verified 2006-02

CONDITIONS: Gastric Variceal Hemorrhage
Keywords: gastric varices; liver cirrhosis; hepatocelluar carcinoma; rebleeding; long-term
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis

INTERVENTIONS:
Procedure: cyanoacrylate injection to treat gastric variceal hemorrhage

SUMMARY:
The purpose of this study was to test the hypothesis by comparing the efficacy of cyanoacrylate injection (GVO) and band ligation (GVL) in the treatment of acute GVH in liver cirrhotic patients with or without concomitant hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Gastric variceal hemorrhage (GVH) has a poorer prognosis than esophageal variceal hemorrhage. However, data on its optimal treatment are limited. We designed a prospective study to compare the efficacy of endoscopic band ligation (GVL) and endoscopic N-butyl-2-cyanoacrylate injection (GVO). Liver cirrhotic patients with or without concomitant hepatocelluar carcinoma (HCC) and patients presenting with acute GVH were randomized into two treatment groups. Forty-eight patients received GVL, and another 49 patients received GVO. Both treatments were equally successful in controlling active bleeding (14/15 vs. 14/15, P = 1.000). More of the patients who underwent GVL had GV rebleeding (GVL vs. GVO, 21/48 vs. 11/49; P = .044). The 2-year and 3-year cumulative rate of GV rebleeding were 63.1% (95% confidence interval [CI], 44.5%-81.7%), 72.3% (95% CI, 51.3%-93.3%) for GVL and 26.8% (95% CI, 12.5%-41.1%), 26.8% (95% CI, 12.5%-41.1%) for GVO; P = .0143, log-rank test. The rebleeding risk of GVL sustained throughout the entire follow-up period. Multivariate Cox regression indicated that concomitance with HCC (relative hazard: 2.453, 95% CI: 1.036-5.806, P = .041) and the treatment method (GVL vs. GVO, relative hazard: 2.660, 95% CI: 1.167-6.061, P = .020) were independent factors predictive of GV rebleeding. There was no difference in survival between the two groups. Severe complications due to these two treatments were rare. In conclusion, the efficacy of GVL to control active GVH appears to have no difference with GVO, but GVO is associated with a lower GV rebleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18 and 80 years and had endoscopy-proven acute gastric variceal hemorrhage (GVH)

Exclusion Criteria:

* Cases with concomitant large GV and large EV, but without stigmata of recent bleeding
* Cases had previous endoscopic, surgical treatment or transjugular intrahepatic portosystemic shunt for GVH
* Cases had a terminal illness of any major organ system, like heart failure, uremia, chronic obstructive pulmonary disease, or nonhepatic malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120

PRIMARY OUTCOMES:
Comparing the efficacy of cyanoacrylate injection (GVO) and band ligation (GVL) in the treatment of acute gastric variceal hemorrhage (GVH) in liver cirrhotic patients

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ming-Chih Hou, M.D., Taipei, Taiwan